CLINICAL TRIAL: NCT02222012
Title: Identification of Neuromarkers in Novel Neuromodulation Treatment in Major Depressive Disorder Based on Integration of Multiple Monitoring Measures
Brief Title: Neuromarkers Identification in Major Depressive Disorder Based on Monitoring Measures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shalvata Mental Health Center (Other)
Collaborators: Beer Yaakov Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: sha-04-14
Record Dates: First submitted 2014-08-17; First posted 2014-08-21 (Estimated); Last update posted 2014-08-21 (Estimated); Status verified 2014-08

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- single channel (Active Comparator)
  Interventions: Device: single channel "Multiway Coil®"
- Two channels "Multiway stimulator coil®" (Brainsway Ltd.) (Experimental)
  Interventions: Device: Two channels "Multiway stimulator coil®" (Brainsway Ltd.)

INTERVENTIONS:
Device: single channel "Multiway Coil®" — During the single channel treatment trial period the patients will receive the following dose of rTMS: 10 Hz - left DLPFC ( 10 Hz, at 120% MT, 3 sec pulse train, 20 second inter-train interval, 55 trains, i.e. a total of 1650 pulses per session, a total of 20 sessions in the study and a cumulative exposure (total number of pulses) of 33,000pulses in 4 weeks).
  Arms: single channel
Device: Two channels "Multiway stimulator coil®" (Brainsway Ltd.) — During the two channels treatment trial period the patients will receive the following dose of rTMS: 10 Hz- left DLPFC, 1Hz - right DLPFC together.
  10 Hz protocol: ( 10 Hz, at 120% MT, 3 sec pulse train, 20 second inter-train interval, 55 trains, i.e. a total of 1650 pulses per session, a total of 20 sessions in the study and a cumulative exposure (total number of pulses) of 33,000pulses in 4 weeks)
  1 Hz protocol:
  1 Hz, at 120% MT, 5 min pulse train, 1 min inter-train interval, 6 trains, i.e. a total of 1800 pulses per session, a total of 20 sessions in the study and a cumulative exposure (total number of pulses) of 36,000 pulses in 4 weeks).
  Arms: Two channels "Multiway stimulator coil®" (Brainsway Ltd.)

SUMMARY:
The investigators propose a multi-source pattern which integrates neuroimaging data associated with multiple, symptom-related neural processes relevant in depression to improve classification accuracy. The investigators conclude that combining brain activation related to the core-symptoms of depression using the multi-source monitoring data substantially increases classification accuracy while providing a sparse relational neuromarkers-model for future prediction.

DETAILED DESCRIPTION:
The "Multiway stimulator coil®" (Brainsway Ltd.) is a novel TMS stimulator with several new and unique properties. Currently standard TMS devices include a single channel, and can operate only a single coil. The "Multiway stimulator coil®" (Brainsway Ltd.) includes two channels which can operate two independent TMS coils, either simultaneously or sequentially.

The "Multiway stimulator coil®" (Brainsway Ltd.) may be used to obtain a differential activation of various brain regions. For instance it can be used to induce high frequency stimulation of a certain brain region, thus inducing facilitation, while simultaneously stimulate at low frequency in another brain region, leading to inhibition.

In the current study the investigators propose a multi-source pattern which integrates neuroimaging data associated with multiple, symptom-related neural processes relevant in depression to improve classification accuracy. The investigators conclude that combining brain activation related to the core-symptoms of depression using the multi-source monitoring data substantially increases classification accuracy while providing a sparse relational neuromarkers-model for future prediction.

The purpose of the study is to to monitor and optimize the anti depressive effect of brain modulation technique using novel multi model monitoring approach.

Subjects will be treated with one of two designs of the study device (the "Multiway Coil®"):

1. Single Channel with a coil placed over the left PFC (10 Hz).
2. Two channels: a. 10 Hz over the left PFC. b. 1 Hz over the right PFC.

All subjects in the current study will undergo monitoring procedure inclusive of functional MRI and electroencephalogram.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient
* Diagnosed by senior psychiatrist as suffering from major depression episode according to DSM IV using the Structured Clinical Interview for DSM-4 (SCID).
* Rating on HDRS-21>20.
* Age: 18-68 years.
* Treated for the current depressive episode, at least four weeks, with at least one antidepressant in accepted dose, without improvement, according to their medical chart and ATHF ( antidepressant treatment history form) instruction guidelines .
* Gave informed consent for participation in the study.
* Negative answers on safety screening questionnaire for transcranial magnetic stimulation.

Exclusion Criteria:

* Diagnosis as suffering from other diagnosis on axis 1 ( like: schizophrenia, bipolar disorder, psychotic depression, geriatric depression).
* Diagnosis as suffering from Severe Borderline Personality Disorder or hospitalized due to exacerbation related to of borderline personality disorder.
* Substantial suicidal risk as judged by the treating psychiatrist.
* Attempted suicide in the past year.
* Any current unstable medical or surgical illness.
* History of seizure or heat convulsion.
* History of epilepsy or seizure in first degree relatives.
* History of head injury.
* History of any metal in the head (outside the mouth).
* Known history of any metallic particles in the eye, implanted cardiac pacemaker or any intracardiac lines, implanted neurostimulators, surgical clips, cochlear implants or any medical pumps.
* History of hearing loss.
* History of drug abuse or alcoholism in the last 6 month.
* Pregnancy or not using a reliable method of birth control.
* Systematic and metabolic unstable disorders.
* Inadequate communication with the patient.
* Under custodial care.
* Participation in current clinical study or clinical study within 30 days prior to this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-08; Primary Completion 2014-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Clinical antidepressant response as defined by decline of HDRS-21 score over time | 20 day
  Clinical antidepressant response at the end of the treatment, defined as a decline in Hamilton depression rating scale (HDRS-21) from the baseline rating by 50%.

SECONDARY OUTCOMES:
Symptomatic improvement | day 20
  Symptomatic improvement at the 4-week end point as measured with Hamilton Anxiety Rating Scale ( HARS)
Clinical antidepressant remission as defined by decline of HDRS-21 score over time | Day 20
  Clinical antidepressant remission at the end of the treatment, defined as exit Hamilton Depression Rating Scale <10.
Symptomatic improvement | day 20
  Symptomatic improvement at the 4-week end point as measured with Quick Inventory of Depressive Symptomatology - Self Report (QIDS-SR)
Symptomatic improvement | day 20
  Symptomatic improvement at the 4-week end point as measured with Clinical Global Impression (CGI)

CONTACTS AND LOCATIONS:
Overall Officials: Yuval Bloch, Md, Phd, Principal Investigator — Shalvata Mental Health Center
Locations (1):
- Shalvata Mental Health Center, Hod HaSharon, Israel